CLINICAL TRIAL: NCT06057870
Title: Feasibility of Wearable Biosensors for Monitoring Daily Activity, Heart Rate, and Sleep Among Patients With Decompensated Cirrhosis
Status: Not yet recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Shelly Lu, Principal Investigator, Cedars-Sinai Medical Center
Other Study IDs: STUDY00002606
Record Dates: First submitted 2023-08-24; First posted 2023-09-28 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Liver Cirrhosis, Alcoholic
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Application on Apple watch — To determine the feasibility and engagement with remote management of acutely decompensated cirrhosis patients using CirrhoCare® App, CyberLiver ART App, and remote monitors by assessing patient adherence to the monitoring device and the Apps over a 3-month period.

SUMMARY:
In this protocol, the investigators will determine compliance, acceptability, and patient satisfaction regarding the use of remote monitors and summarize changes in activity over time among patients with decompensated cirrhosis.

This is a feasibility pilot study that will recruit 20 patients. The investigators plan to determine the feasibility of wearable devices to remotely monitor daily activity (e.g., physical activity, sedentary time, sleep), cognitive function, blood pressure, and weight in patients with decompensated cirrhosis, by assessing patient compliance. A patient is considered compliant if they wear the wristwatch at least 10 hours per day and use the Apps, body weight scale, and blood pressure monitor for at least 4 of 7 days

ELIGIBILITY:
Inclusion Criteria:

- Patients with an admission diagnosis of decompensated cirrhosis based on Child-Turcotte-Pugh score of ≥ 7 or MELD-Na score ≥ 15, measured prior to discharge from the hospital. Cirrhosis of any etiology may be included. However, patients with cirrhosis due to autoimmune hepatitis must be on a stable corticosteroid dose for three months or more before study inclusion.

2.4.2 18 years or older 2.4.3 Ambulatory (use of walking aids, such as cane and rollator, is acceptable) 2.4.4 Have an understanding, ability, and willingness to fully comply with study procedures and restrictions as determined by the principal investigator.

2.4.5 Informed consent obtained from the subject and the ability of the subject to comply with the requirements of the study.

Exclusion Criteria:

* 2.5.1 Using a pacemaker, implantable cardiac defibrillator, neurostimulator, implantable hearing aids, cochlear implants, or other electronic medical equipment. However, removable hearing aids are permitted.

2.5.2 Presence of advanced or terminal stage hepatocellular carcinoma 2.5.3 Patients with current extrahepatic malignancies including solid tumors and hematologic disorders 2.5.4 Patients with an ongoing ACLF (see diagnostic criteria in reference16) 2.5.5 Patients with a history of significant extrahepatic disease with impaired short-term prognosis, including congestive heart failure New York Heart Association Grade III/IV, COPD GOLD >2, chronic kidney disease defined by KDIGO criteria, or under renal replacement therapy.

2.5.6 Presence of any extra-hepatic malignancy not in remission for > 12 months 2.5.7 Pregnancy, since being pregnant may alter heart rate and sleep patterns. Women of childbearing age remain eligible.

2.5.8 Inability or refusal to provide informed consent by the patient 2.5.9 Patients with hepatic encephalopathy New Haven grade 1 or greater. 2.5.10 Any records flagged "break the glass" or "research opt out."

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with decompensated cirrhosis who are admitted to the hospital will be screened for eligibility and approached before discharge. If they are eligible for the study and if so, the potential subject is presented with an option of enrolling.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of using remote health monitoring | up to 1 year
  To determine the feasibility and engagement with remote management of acutely decompensated cirrhosis patients using CirrhoCare® App, CyberLiver ART App, and remote monitors by assessing patient adherence to the monitoring device and the Apps over a 3-month period. After the 3-month study period, the participants can opt to remain in contact using the App. If they agree, they will be contacted at 6 months and a year.